CLINICAL TRIAL: NCT02860689
Title: Predictive Factors for Male Sexual Dysfunction After Traumatic Spinal Cord Injury
Status: Completed | Type: Observational
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Josepha Karinne de Oliveira Ferro, Physical Therapist, Universidade Federal de Pernambuco
Other Study IDs: Spinal Cord 2016
Record Dates: First submitted 2016-07-31; First posted 2016-08-09 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Male Sexual Dysfunction; Spinal Cord Injury
Keywords: Sexuality; Spinal cord injuries; Penile erection; erectile dysfunction; Psychological Sexual Dysfunctions
MeSH Terms: conditions — Spinal Cord Injuries; Sexuality; Erectile Dysfunction; Sexual Dysfunctions, Psychological

STUDY DESIGN:
Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: using questionnaires - International Index Erectile Function — using questionnaires

SUMMARY:
Objective: To analyze the association between sexual function of men with spinal cord injury with possible predictive factors for dysfunction.

DETAILED DESCRIPTION:
Method: Observational study (CAAE 41221414.5.0000.5208) conducted with 45 men, mean age 34 (CI 31.5 to 37.1), with spinal cord injury and active sex life. Sexual function was assessed by the International Index of Erectile Function and level and degree of injury were determined following the guidelines of the International Standards for Neurological and Functional Examination Classification of Spinal Cord Injury. Descriptive statistical techniques were applied and multivariate analysis using logistic regression adjusted to observe the association between factors, with 0.05 significance level.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of traumatic spinal cord injury, injury time less than six months heterosexual and sexually active

Exclusion Criteria:

* patients who had erectile dysfunction attributed to endocrine or metabolic disease order, those who underwent surgery in the genital area, such as radical prostatectomy or penile implant and cognitive impairment

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study included 45 men, aged between 18 and 60 years with a clinical diagnosis of traumatic spinal cord injury, injury time less than six months heterosexual and sexually active. The study excluded patients who had erectile dysfunction attributed to endocrine or metabolic disease order, those who underwent surgery in the genital area, such as radical prostatectomy or penile implant and cognitive impairment.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2015-03; Primary Completion 2016-01 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Male Sexual Dysfunction | one day
  Male Sexual Dysfunction assessed by International Index of Erectile Function (IIEF)

SECONDARY OUTCOMES:
Level of neurological lesion | one day
  Level of neurological lesion assessed by ASIA Impairment Scale (AIS) according to the International Standards for Neurological and Functional Examination Classification of Spinal Cord Injury
Degree of neurological lesion | one day
  Degree of neurological lesion assessed by ASIA Impairment Scale (AIS) according to the International Standards for Neurological and Functional Examination Classification of Spinal Cord Injury
Depression | one day
  Depression assessed by Beck Depression Inventary (BDI)

CONTACTS AND LOCATIONS:
Overall Officials: Josepha KO Ferro, master, Principal Investigator — Universidade Federal de Pernambuco
Locations (1):
- Josepha Karinne de Oliveira Ferro, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: No